CLINICAL TRIAL: NCT05274763
Title: A Feasibility Study of Chaplain-Delivered Compassion Meditation for Patients Receiving Stem Cell Transplantation
Brief Title: Chaplain-Delivered Compassion Meditation to Improve Quality of Life in Patients Receiving a Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Mascaro, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003563; NCI-2022-00233 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00003563; EU5492-21 (Other: Emory University Hospital/Winship Cancer Institute); K01AT010488 (NIH); P30CA138292 (NIH)
Record Dates: First submitted 2022-02-25; First posted 2022-03-10 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma; Plasma Cell Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Spiritual Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Experimental): Patients undergo 4 to 8 sessions (2-4 per week) of Compassion Centered Spiritual Health (CCSH) over 30 minutes with a chaplain while impatient.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Spiritual Therapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Spiritual Therapy — Deliver or undergo Compassion Centered Spiritual Health (CCSH) session

SUMMARY:
This clinical trial tests whether chaplain-delivered compassion centered spiritual health (CCSH) works to improve quality of life in patients receiving a stem cell transplant. Compassion Centered Spiritual Health (CCSH) is a secularized, research-based mindfulness and compassion meditation program designed to expand and strengthen compassion for self and others. Practices include training in attentional stability and increased emotional awareness, as well as targeted reflections to appreciate one's relationship with self and others. By centering the mind, controlling negative thoughts, and cultivating personal resiliency and an inclusive and more accurate understanding of others, Compassion Centered Spiritual Health (CCSH) may help improve response to stress and reduce inflammation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the feasibility, adoption, extent of implementation, and fidelity of chaplain-delivered Compassion Centered Spiritual Health (CCSH).

OUTLINE:

Patients undergo 4 to 8 sessions (2-4 per week) of Compassion Centered Spiritual Health (CCSH) over 30 minutes with a chaplain while impatient.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Within 6 weeks of scheduled hematopoietic stem cell transplant (HSCT)
* PATIENT: > 18 years of age
* PATIENT: Speak and read English
* CHAPLAIN: Emory Healthcare Chaplain

Exclusion Criteria:

* CHAPLAIN: There will be no exclusion criteria and no consequence to the chaplains for refusing to volunteer
* PATIENT: Neurologic or cognitive problems that preclude chaplain-delivered Compassion Centered Spiritual Health (CCSH)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mascaro, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Supportive Care: Compassion Centered Spiritual Health (CCSH): Patients undergo 4 to 8 sessions (2-4 per week) of Compassion Centered Spiritual Health (CCSH) over 30 minutes with a chaplain while impatient.
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Spiritual Therapy: Deliver or undergo Compassion Centered Spiritual Health ssession
Period: Overall Study
Arm/Group | Supportive Care: Compassion Centered Spiritual Health (CCSH)
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Supportive Care (CCSH): Patients undergo 4 to 8 sessions (2-4 per week) of CCSH over 30 minutes with a chaplain while impatient.
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Spiritual Therapy: Deliver or undergo CCSH session
Arm/Group | Supportive Care (CCSH)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 57 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Fidelity to Intervention Delivery
Description: Chaplains will deliver between four and eight 30-minute sessions (2-4 times per week) to evaluate the fidelity of implementation (FOI).
  Administer the (4 min) Scottish Patient Reported Outcome Measure. The Patient Reported Outcome Measure is an 18-item Likert-scale that assesses how a hospitalized patient felt about the pastoral care visit both during the consult and after it.
  The scale will indicate the following range: 5-25, with higher scores indicating more improvement as a result of the chaplain visit and lower scores indicating less improvement as a result of the chaplain visit.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Supportive Care: Compassion Centered Spiritual Health (CCSH): Patients undergo 4 to 8 sessions (2-4 per week) of Compassion Centered Spiritual Health over 30 minutes with a chaplain while impatient.
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Spiritual Therapy: Deliver or undergo Compassion Centered Spiritual Health session
Arm/Group | Supportive Care: Compassion Centered Spiritual Health (CCSH)
Number analyzed (Participants) | 30
score on a scale | 19.9 (4.84)

2. Secondary Outcome: Number of Sessions Completed
Description: Adherence will be evaluated as the percent of sessions completed by patients and characterized as "low" (< 70%), "moderate" (70-80%),"high" (> 80%) adherence.
Time Frame: Up to 3 months
Population: Evaluated the number of participants categorized as low (< 70%), medium (70 - 80%) and high (> 80%) adherence.
Measure: Count of Participants; unit: Participants
Groups:
- Supportive Care Compassion Centered Spiritual Health (CCSH): Patients undergo 4 to 8 sessions (2-4 per week) of Compassion Centered Spiritual Health over 30 minutes with a chaplain while impatient.
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Spiritual Therapy: Deliver or undergo Compassion Centered Spiritual Health session
Arm/Group | Supportive Care Compassion Centered Spiritual Health (CCSH)
Number analyzed (Participants) | 30
Participants
  Low: participants who had low adherence range | 12
  Medium: participants who had medium adherence | 10
  High: participants who had high adherence | 8

3. Secondary Outcome: Percentage of Cognitive Based Compassion Training
Description: Dosage is quantified as the amount (percentage) of cognitive based compassion training (CBCT) that patients receive. Characterize the modal number of sessions received as well as the range of sessions completed by all patients. From the range, sessions will be categorized of "low" (<70%), "moderate" (70-80%),"high" (> 80%) dosage.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care: Compassion Centered Spiritual Health (CCSH)
Number analyzed (Participants) | 30
Participants
  Number of participants enrolled who did not complete any sessions | 3
  Number of Enrolled Participants that Completed a Single Session | 9
  Number of Enrolled Participants that Completed Two Sessions | 10
  Number of Enrolled Participants that Completed Three Sessions | 3
  Number of Enrolled Participants that Completed Four Sessions | 4
  Number of Enrolled Participants that Completed Five Sessions | 1
  Number of Enrolled Enrolled Participants with High Dosage to CCSH | 8
  Number of Enrolled Participants with Moderate Dosage to CCSH | 10
  Number of Enrolled Participants with Low Dosage to CCSH | 12

4. Secondary Outcome: Responsiveness
Description: Evaluate the rate of responsiveness in each session, operationalized as "maximally," "moderately", or "minimally" enthusiastic and attentive during each.
Time Frame: Up to 3 months
Population: The 30 participants' responsiveness was rated for 54 sessions
Measure: Number; unit: number of sessions
Arm/Group | Supportive Care Compassion Centered Spiritual Health (CCSH)
Number analyzed (Participants) | 30
number of sessions
  Number of sessions rated as maximum responsiveness | 33
  Number of sessions rated as moderate Responsiveness | 17
  Number of sessions rated as minimal Responsiveness | 4

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: No adverse event was reported.
Arm/Group | Supportive Care (CCSH)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
This study was not designed to evaluate efficacy, therefore no statistical analysis was developed or associated with this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT05274763/Prot_000.pdf
  • Informed Consent Form (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT05274763/ICF_001.pdf